CLINICAL TRIAL: NCT04350632
Title: Reproducibility of External Anal Sphincter Elastic Properties Assessment Using Elastography During Pregnancy
Acronym: SEA ELASTO 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A00762-37
Record Dates: First submitted 2020-04-07; First posted 2020-04-17 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Obstetric Anal Sphincter Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Shear wave elastography assessment of the external anal sphincter — Assessment of the external anal sphincter viscoelastic properties using shear wave elastography technology
  * Women in lithotomy position with an empty bladder
  * The linear probe is applied on transversal plane on the perineal with a transperineal approach
  * The external anal sphincter will be identified in 2D ultrasound using a SL 18-5 linear probe
  * Viscoelastic properties of the muscle will be assessed by measuring the shear modulus at rest, Valsalva maneuver and contraction
  * Exactly the same investigations will be performed for the two visits planned in the protocol. In the first visit, it will be one single observer and for the second it will be 2 observers.
  * Data about the mode of delivery and the occurrence of OASI will be collected into women's medical fil

SUMMARY:
The risk prediction of obstetric anal sphincter injury couyl be optimized by considering pregnant women's anal sphincter intrinsic viscoelastic properties. Shear wave elastography is a new technology that allowed an in vivo assessment of viscoelastic properties of tissues such as muscles. The main endpoint of this study is to assess the intra-observer and the inter-observer reproducibility of a the external anal sphincter assessment using shear wave elastography in term pregnant women.

DETAILED DESCRIPTION:
Investigations Assessment of the external anal sphincter viscoelastic properties using shear wave elastography technology using a transperineal approach in term pregnant women in two visits (the 1st one with only one observer and the second one with two observers)

Follow up Prospective study including nulliparous term pregnant women with 2 visits planned, spaced at least by 12 hours and, for the most, 7 days.

Primary outcome: The mean value of shear modulus measures in the external anal sphincter for the three considered conditions (rest, Valsalva maneuver and contraction) at each visit and for each observer with a calculation of Intraclass Correlation Coefficient and Variation Coefficient.

Secondary outcomes: The secondary outcomes will be the percentage of completed procedure (ability to see the external sphincter and to obtain a measure of the shear modulus), the existence of a perineal tear according the RCOG-OMS classification and the answer to an acceptability question.

Study design: Prospective monocentric study including nulliparous term pregnant women with two visits spaced of at least 12 hours and, for the most, 7 days.

Interventions: Assessment of the external anal sphincter viscoelastic properties using shear wave elastography technology

* Women in lithotomy position with an empty bladder
* The linear probe is applied on transversal plane on the perineal with a transperineal approach
* The external anal sphincter will be identified in 2D ultrasound using a SL 18-5 linear probe
* Viscoelastic properties of the muscle will be assessed by measuring the shear modulus at rest, Valsalva maneuver and contraction
* Exactly the same investigations will be performed for the two visits planned in the protocol. In the first visit, it will be one single observer and for the second it will be 2 observers.
* Data about the mode of delivery and the occurrence of OASI will be collected into women's medical file

Number of subjects: 40 volunteers pregnant women are planned for this research

Statistical analysis: The number of successful procedures will be reported as effectives and percentages.

Reproducibility will be reported by calculating the coefficient of variation and the intraclass correlation coefficient. The level of significance will be considered for p<0.05

Conditions : Obstetric anal sphincter injury

Keywords: OASI; childbirth; perineal traumatism; delivery; biomechanics; shear wave elastography

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged of 18 years or more
* 37 weeks or more of pregnancy
* without any previous delivery (vaginal or cesarean delivery)
* body mass index < 35Kg.m-2
* without history of Crohn's disease
* without history of peri anal surgery
* without any proctologic disease
* without any muscular chronic disease
* having a normal pregnancy
* without any untreated psychiatric disorders
* without any judicial protection
* affiliated to a health insurance

Exclusion Criteria:

* pregnant women younger than 18 years old
* obstetric term inferior than 37 weeks
* history of vaginal and/or cesarean delivery
* body mass index of 35Kg.m-2 or more
* history of Crohn's disease
* history of peri anal surgery
* proctologic disease
* muscular chronic disease
* pathological pregnancy (intrauterine growth restriction, pre eclampsia etc..)
* untreated psychiatric disorders
* women under judicial protection
* women without affiliated to a health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — obsterics
Enrollment: 40 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-10-07 (Estimated); Study Completion 2021-10-14 (Estimated)

PRIMARY OUTCOMES:
value of shear modulus measures in the external anal sphincter for each visit with the calculation of the ICC | up to seven days
  The mean value of shear modulus measures in the external anal sphincter for the three considered conditions (rest, Valsalva maneuver and contraction) at each visit and for each observer with a calculation of Intraclass Correlation Coefficient
value of shear modulus measures in the external anal sphincter for each visit with the calculation of the coefficent of variation | up to seven days
  The mean value of shear modulus measures in the external anal sphincter for the three considered conditions (rest, Valsalva maneuver and contraction) at each visit and for each observer with a calculation of Variation Coefficient

SECONDARY OUTCOMES:
Perineal tears at childbirth | up to 4 weeks
  the existence of a perineal tear according the RCOG-OMS classification
Feasibility of the assessment of the external anal sphincter: percentage of completed procedure | up to seven days
  percentage of completed procedure (ability to identify the extarnal anal sphincter and to perform a shear wave elastography assessment)
Acceptability of the procedure: question with a scale | up to seven days
  answer to the acceptability question with a scale from 0 to ten

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided